CLINICAL TRIAL: NCT01170182
Title: A Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover Bioequivalence Study to Compare Omeprazole 40 mg DR Capsules Dr. Reddy's Laboratories Ltd.,With Prilosec® 40 mg Merck & Co., Inc.,USA Under Fed Condition
Brief Title: Omeprazole Delayed Release (DR) Capsules Bioequivalence Study of Dr. Reddys Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Assistant Manager - Research & Development, Dr. Reddy's Laboratories Limited,
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7577/05-06
Record Dates: First submitted 2010-05-31; First posted 2010-07-27 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole (Experimental): Omeprazole Delayed Release Capsules of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Omeprazole
- Prilosec (Active Comparator): Prilosec® 40 mg Merck & Co. Inc
  Interventions: Device: Prilosec® 40 mg

INTERVENTIONS:
Drug: Omeprazole — Omeprazole Delayed Release Capsules 40 mg
  Other Names: Prelosec 40 mg
  Arms: Omeprazole
Device: Prilosec® 40 mg — Prilosec® 40 mg
  Other Names: Omeprazole
  Arms: Prilosec

SUMMARY:
This study examines the bioequivalence of Dr. Reddy's Omeprazole delayed release capsules under fed condition.

DETAILED DESCRIPTION:
This is a randomized, two-treatment, two-period, two-sequence, single dose, crossover bioequivalence study to compare Omeprazole 40 mg Delayed Release Capsules (Dr. Reddy's Laboratories Ltd.,) with Prilosec® 40 mg (Omeprazole Delayed Release Capsules) (manufactured by Merck & Co., Inc., USA) in 54 healthy, adult, human subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provided written informed consent.
* Subjects who were healthy within 18-45 years of age, weighing at least 50 kg.
* Body mass index of ≥18 kglm2 and ≤ 25 kg/m2, with body weight not less than 50 kg.
* Subjects with normal health as determined by medical history and physical examination performed within 15 days prior to the commencement of the study (dosing in period-I).
* Subjects with normal ECG, chest X-ray (PA view) and vital signs.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2006-02; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Bose, Dr., Principal Investigator — Vimta Labs Limited, 142, IDA, Phase-II, Cherlapally, Hyderabad, India-500 051